CLINICAL TRIAL: NCT00079183
Title: A Phase II Clinical Trial to Evaluate the Safety and Efficacy of Sirolimus for Secondary Treatment of Chronic Graft-versus-Host Disease
Brief Title: Sirolimus as Secondary Therapy in Chronic Graft-Versus-Host Disease Not Responding To Prior Treatment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Paul Carpenter, Principal Investigator, Fred Hutchinson Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 1706.00; NCI-2011-01817 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2004-03-08; First posted 2004-03-10 (Estimated); Results first posted 2017-05-12 (Actual); Last update posted 2017-06-20 (Actual); Status verified 2017-05

CONDITIONS: Graft Versus Host Disease
MeSH Terms: conditions — Graft vs Host Disease | interventions — Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sirolimus (Experimental): Study participants receive sirolimus added once daily to their baseline combination therapy of prednisone plus either cyclosporine or tacrolimus at the discretion of the managing physician. Treatment other than cyclosporine (or tacrolimus) and prednisone must be discontinued when administration of sirolimus is started. Topical therapy, including psoralen and UVA irradiation (PUVA), glucocorticoid creams, topical tacrolimus, oral beclomethasone, topical azathioprine and ophthalmic glucocorticoids may be given at the discretion of the managing physician in consultation with the transplant center.
  Interventions: Drug: sirolimus

INTERVENTIONS:
Drug: sirolimus — Given PO
  Other Names: AY 22989; Rapamune; rapamycin; SLM

SUMMARY:
This phase II trial studies the side effects and how well sirolimus works as secondary therapy in treating patients with chronic graft-versus-host disease (GVHD) that did not respond to prior treatment. Sirolimus may be an effective treatment for chronic GVHD

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the safety of sirolimus administered at a dose which provides steady-state, whole blood trough levels of 5-10 ng/mL in patients with chronic GVHD.

II. To determine whether administration of sirolimus provides benefit for patients with chronic GVHD that has not responded adequately to previous systemic treatment.

OUTLINE:

Patients receive sirolimus orally (PO) once daily (QD). Patients continue to receive prednisone and cyclosporine or tacrolimus at the discretion of the managing physician.

After completion of study treatment, patients are followed up periodically.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy-confirmed diagnosis of clinical extensive chronic GVHD with inadequate response to previous treatment and where secondary systemic therapy is indicated because of

  * Clinical progression of signs and symptoms of chronic GVHD in a previously involved organ, or
  * Development of signs and symptoms of chronic GVHD in a previously uninvolved organ, or
  * Absence of improvement after 3 months of primary treatment, or
  * Continued need for treatment with prednisone at doses >= 1.0 mg/kg/day for more than 2 months, without qualification for type of donor, graft or conditioning regimen
* Patient or guardian able and willing to provide informed consent
* Stated willingness to use contraception in women of child-bearing potential (Food and Drug Administration [FDA] requirement)
* Stated willingness of the patient to comply with study procedures and reporting requirements
* Stated willingness of the physician most involved in management of chronic GVHD (the "managing physician,") to comply with study procedures and reporting requirements

Exclusion Criteria:

* Fungal or viral infection with no radiographic evidence of improvement during continued appropriate antimicrobial therapy
* Cytomegalovirus (CMV) antigenemia unresponsive to antiviral therapy
* Active disseminated varicella zoster virus (VZV) infection with persistent non-crusted lesions
* Inability to tolerate oral medications
* Absolute neutrophil count (ANC) < 1500/uL
* Platelet count < 50,000/uL
* Persistent or recurrent malignancy, including histopathologic evidence of myeloma or lymphoma; patients with breakpoint cluster region-abelson (bcr/abl) detected by polymerase chain reaction (PCR) assay as the only evidence of persistent chronic myeloid leukemia may be enrolled
* Pregnancy
* Known history of hypersensitivity to sirolimus

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2002-04; Primary Completion 2009-07 (Actual); Study Completion 2010-06-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Carpenter, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (1):
- Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sirolimus
Started | 44
Drop Outs | 7
Completed | 37
Not Completed | 7
Not completed — Withdrawal by Subject | 4
Not completed — Study medication non-compliance | 2
Not completed — Specimen collection non-compliance | 1

BASELINE CHARACTERISTICS:
Population: This includes all 44 consented subjects.
Arm/Group | Sirolimus
Number analyzed (Participants) | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 14
  Between 18 and 65 years | 26
  >=65 years | 4
Age, Continuous [Median (Full Range); unit: years] | 40.55 [1.4 to 72.4]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 42
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 39
  More than one race | 2
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 44

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing Treatment Success
Description: Defined as the absence of any immunosuppressive treatment, including sirolimus, with resolution of all reversible manifestations of chronic GVHD and no additional systemic therapy.
Time Frame: Approximately 7 years
Measure: Count of Participants; unit: Participants
Arm/Group | Sirolimus
Number analyzed (Participants) | 44
Participants | 8

2. Primary Outcome: Number of Participants Experiencing Treatment Failure
Description: Defined as the initiation of additional systemic therapy, development of bronchiolitis obliterans, or death from causes other than recurrent malignancy during primary treatment for chronic GVHD, whichever occurs first.
Time Frame: Approximately 7 years
Measure: Count of Participants; unit: Participants
Arm/Group | Sirolimus
Number analyzed (Participants) | 44
Participants | 9

3. Primary Outcome: Number of Participants Needing Additional Systemic Therapy
Description: Includes any intervention intended to control chronic GVHD through an immunosuppressive effect from oral or parenteral administration of any systemic medication not originally given under auspices of this protocol.
Time Frame: Approximately 7 years
Measure: Count of Participants; unit: Participants
Groups:
- Sirolimus: Study participants receive sirolimus added once daily to their baseline combination therapy of prednisone plus either cyclosporine or tacrolimus at the discretion of the managing physician. Treatment other than cyclosporine (or tacrolimus) and prednisone must be discontinued when administration of sirolimus is started. Topical therapy, including psoralen and UVA irradiation (PUVA), glucocorticoid creams, topical tacrolimus, oral beclomethasone, topical azathioprine and ophthalmic glucocorticoids may be given at the discretion of the managing physician in consultation with the transplant center.
  sirolimus: Given PO
  questionnaire administration: Ancillary studies
  quality-of-life assessment: Ancillary studies
Arm/Group | Sirolimus
Number analyzed (Participants) | 44
Participants
  No additional therapy (off immunosuppressive Rx) | 8
  Additional immunosuppressive therapy (IST) added | 9
  Still on IST but no new IST added | 27

4. Primary Outcome: Number of Participants With Recurrent Malignancy
Description: Defined as clinical or histopathologic evidence demonstrating the presence of any malignancy considered as the indication for transplant. Recurrent malignancy will also be defined as any post-transplant intervention not routinely used to prevent the development of overt recurrence, prompted by laboratory evidence of persisting malignant cells but without clinical or histopathologic evidence of recurrence.
Time Frame: Approximately 7 years
Measure: Count of Participants; unit: Participants
Arm/Group | Sirolimus
Number analyzed (Participants) | 44
Participants | 5

5. Secondary Outcome: Proportion of Patients Who Discontinue Administration of Sirolimus Because of Toxicity
Time Frame: Approximately 7 years
Measure: Count of Participants; unit: Participants
Arm/Group | Sirolimus
Number analyzed (Participants) | 44
Participants | 6

6. Secondary Outcome: Proportion With Infections Categorized by Organism
Time Frame: Approximately 7 years
Measure: Count of Participants; unit: Participants
Arm/Group | Sirolimus
Number analyzed (Participants) | 44
Participants
  Proportion of pts with at least 1 infection | 21
  Proportion of pts with at least 1 bacterial inf'n | 19
  Proportion of pts with at least 1 viral inf'n | 6
  Proportion of pts with at least 1 fungal inf'n | 4
  Proportion of pts with culture negative sepsis | 1

7. Secondary Outcome: Secondary Malignancies
Description: Proportion of participants who developed at least one secondary malignancy by 7 years
Time Frame: Up to 7 years
Measure: Count of Participants; unit: Participants
Arm/Group | Sirolimus
Number analyzed (Participants) | 44
Participants
  Proportion with any second malignancy | 15
  Proportion with any subsequent skin malignancy | 13
  Proportion with subsequent oral malignancy | 3
  Prop'n with subsequent prostate adenocarcinoma | 1
  Prop'n with subsequent renal cell carcinoma | 1
  Proportion with subsequent bladder carcinoma | 1
  Prop'n with post-BMT lymphoproliferative disease | 1

8. Secondary Outcome: Duration of Treatment With Prednisone
Time Frame: Approximately 7 years
Measure: Mean (Full Range); unit: Months
Arm/Group | Sirolimus
Number analyzed (Participants) | 44
Months | 45 [3 to 54]

9. Secondary Outcome: Probability of Survival Without Recurrent Malignancy
Description: Kaplan-Meier estimate assessed at 7 years for probability of survival without recurrent malignancy.
Time Frame: Approximately 7 years
Measure: Number (95% Confidence Interval); unit: disease free survival probability
Arm/Group | Sirolimus
Number analyzed (Participants) | 44
disease free survival probability | 0.54 [0.41 to 0.71]

10. Secondary Outcome: Probability of Overall Survival
Description: Kaplan-Meier estimate assessed at 7 years
Time Frame: Approximately 7 years
Measure: Number (95% Confidence Interval); unit: survival probability
Arm/Group | Sirolimus
Number analyzed (Participants) | 44
survival probability | 0.59 [0.46 to 0.75]

11. Secondary Outcome: Probability of Cumulative Incidence of Death Without Recurrent Malignancy
Description: Analyzed with recurrent malignancy as a competing risk factor. Assessed at 7 years.
Time Frame: Approximately 7 years
Measure: Number (95% Confidence Interval); unit: probability
Arm/Group | Sirolimus
Number analyzed (Participants) | 44
probability | 0.25 [0.13 to 0.39]

12. Secondary Outcome: Probability of Cumulative Incidence of Recurrent Malignancy
Description: Analyzed with death as a competing risk factor. Assessed at 7 years.
Time Frame: Approximately 7 years
Measure: Number (95% Confidence Interval); unit: probability
Arm/Group | Sirolimus
Number analyzed (Participants) | 44
probability | 0.20 [0.10 to 0.33]

ADVERSE EVENTS:
Arm/Group | Sirolimus
All-Cause Mortality (participants affected / at risk) | 15/44
Serious Adverse Events (participants affected / at risk) | 22/44
Other Adverse Events (participants affected / at risk) | 30/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sirolimus (N=44)
Hospitalized for Congestive Heart Failure (Cardiac disorders) | 1 (1)
Hospitalized for Chest Pain (Cardiac disorders) | 1 (1)
Hospitalized for Deep Vein Thrombosis (DVT) (Blood and lymphatic system disorders) | 2 (2)
Hospitalized for Hemolytic-uremic syndrome (HUS) (Blood and lymphatic system disorders) | 2 (2)
Hospitalized for Hypertension (Cardiac disorders) | 1 (1)
Hospitalized for Thrombotic Thrombocytopenic Purpura(TTP) (Blood and lymphatic system disorders) | 1 (1)
Hospitalized for Idiopathic Thrombocytopenic Purpura (ITP) (Blood and lymphatic system disorders) | 1 (1)
Hospitalized for Fever (Infections and infestations) | 1 (1)
Hospitalized for Fatigue (General disorders) | 1 (1)
Hospitalized for Dizziness (Nervous system disorders) | 1 (1)
Hospitalized for Dehydration (Gastrointestinal disorders) | 3 (3)
Hospitalized for Refractory Diarrhea (Gastrointestinal disorders) | 1 (1)
Hospitalized for GVHD Flare (Surgical and medical procedures) | 3 (3) — Graft vs. Host Disease
Hospitalized for Vitamin K Deficiency (Immune system disorders) | 1 (1)
Hospitalized for CMV (Cytomegalovirus Colitis) Enteritis (Infections and infestations) | 1 (1)
Hospitalized for Coag Negative Staph Bacteremia (Infections and infestations) | 3 (3)
Hospitalized for Pneumonia (Infections and infestations) | 10 (10)
Hospitalized for Enterobacter Bacteremia (Infections and infestations) | 3 (3)
Hospitalized for Pseudomonas Aeruginosa Bacteremia (Infections and infestations) | 1 (1)
Hospitalized for Streptococcus Viridans Bacteremia (Infections and infestations) | 2 (2)
Hospitalization for Candida Parapsilosis (Infections and infestations) | 1 (1)
Hospitalized for Septic Shock (Infections and infestations) | 1 (1)
Hospitalized for Hyperglycemia (Endocrine disorders) | 1 (1)
Hospitalized for Sinusitis (Infections and infestations) | 3 (4)
Hospitalized for Anorexia (Gastrointestinal disorders) | 1 (1)
Hospitalized for Otitis Media (Ear and labyrinth disorders) | 1 (1)
Hospitalized for Renal Insufficiency (Renal and urinary disorders) | 4 (4)
Hospitalized for C. Difficile (Infections and infestations) | 1 (1)
Hospitalized for Parainfluenza (Infections and infestations) | 1 (1)
Hospitalization for Respiratory Syncytial Virus (Infections and infestations) | 2 (2)
Hospitalization for Chicken Pox (Infections and infestations) | 1 (1)
Hospitalization for Staphylococcus aureus (Infections and infestations) | 1 (1)
Hospitalization for CMV Mucositis (Infections and infestations) | 1 (1)
Hospitalization for Haemophilus influenzae (Infections and infestations) | 1 (1)
Hospitalization for Staphylococcus epidermidis (Infections and infestations) | 1 (1)
Hospitalization for Micrococcus bacteremia (Infections and infestations) | 1 (1)
Hospitalization for Staphylococcus Hickman Site Infection (Infections and infestations) | 1 (1)
Hospitalization for Hip Replacement (Musculoskeletal and connective tissue disorders) | 1 (2) — First event was total right hip replacement due to AVN steroid use. Second event was total left hip replacement due to AVN steroid use
Hospitalized for Chylothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hospitalized for Oliguric Failure (Renal and urinary disorders) | 1 (1)
Hospitalized for tumor in back (relapse) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Hospitalized for Pancytopenia (Blood and lymphatic system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sirolimus (N=44)
Neutropenia (Blood and lymphatic system disorders) | 4 (6)
Anemia (Blood and lymphatic system disorders) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 4 (4)
Hypertension (Cardiac disorders) | 4 (4)
Fatigue (General disorders) | 1 (1)
Diabetic Foot Ulcers (Endocrine disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 5 (6)
Nausea (Gastrointestinal disorders) | 3 (3)
Vomiting (Gastrointestinal disorders) | 3 (3)
Bronchitis (Infections and infestations) | 3 (3)
Pneumonia (Infections and infestations) | 2 (3)
C. Difficile (Infections and infestations) | 2 (3)
Shingles (Infections and infestations) | 1 (1)
sinusitis (Infections and infestations) | 5 (5)
Otitis Media (Infections and infestations) | 2 (3)
Chicken Pox (Infections and infestations) | 1 (1)
Strep Throat (Infections and infestations) | 2 (2)
Eye Infection (Eye disorders) | 2 (2)
Coag Negative Staph (Infections and infestations) | 1 (1)
Left Parotid Gland Infection (Infections and infestations) | 1 (1)
Pseudomonas aeruginosa (Infections and infestations) | 1 (1)
Aspergillus (Infections and infestations) | 1 (1)
BK Virus (Infections and infestations) | 1 (1)
Lower Extremity Edema (Skin and subcutaneous tissue disorders) | 12 (12)
Hyperlipidemia (Metabolism and nutrition disorders) | 11 (12)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 3 (3)
Depression (Nervous system disorders) | 4 (4)
Renal Insufficiency (Renal and urinary disorders) | 10 (12)
Basal and Squamous Cell (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (5)
Urinary Bladder Tumor (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes